CLINICAL TRIAL: NCT01230034
Title: Randomized, Controlled, PROBE Trial, Evaluating the Antiproteinuric Effect of Imidapril Versus Ramipril in Type 2 Diabetic Patients and Mild to Moderate Hypertension With Microalbuminuria
Brief Title: Antiproteinuric Effect of Imidapril Versus Ramipril in Type 2 Diabetic and Hypertensive Patients With Microalbuminuria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Prof. GianMario Frigo, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV001DIM2010; 2010-023332-17 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus; Microalbuminuria
Keywords: Imidapril, Ramipril, Hypertension, Type 2 diabetes mellitus, Microalbuminuria
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Ramipril; imidapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imidapril (Experimental): 10 and 20 mg/day, pill
  Interventions: Drug: Imidapril
- Ramipril (Active Comparator): 5 and 10 mg/day, pill
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — pill, 5 and 10 mg/day, od, 24 weeks
  Arms: Ramipril
Drug: Imidapril — pill, 10 and 20 mg/day, od, 24 weeks
  Arms: Imidapril

SUMMARY:
Numerous clinical and experimental data show that the elective treatment of diabetic nephropathy should be based on drugs that inhibit the renin-angiotensin system (RAS). Albuminuria is a marker of risk not only renal but also cardiovascular and diabetic patients with concomitant non-diabetic nephropathy, on the other hand, drugs blocking the renin-angiotensin system available so far, namely ACE inhibitors and angiotensin antagonists II have proven effective in reducing proteinuria in power even if different therapeutic drug to drug. ACE inhibitors are one of the most known and used treatment options for blocking the renin-angiotensin system in patients with microalbuminuria. Drugs such as enalapril, lisinopril and ramipril are standard therapy in diabetic patients with micro or macroalbuminuria. However, it is still unclear whether their efficacy is, from this point of view, the same or varies from drug to drug. This is particularly true in the diabetic microalbuminuria, a condition in which there is sufficient documentation to prove that ramipril is effective. The main objective of this study was to assess the magnitude and trend of the time and to the antiproteinuric effect of antihypertensive 10-20mg/die imidapril versus ramipril 5-10 mg / day in hypertensive patients with type 2 diabetes and microalbuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure> 130/80 ≤ 170/100 mmHg at the end of the period of wash-out
* Type 2 diabetes mellitus well controlled by medication and / or compliance with diet (HbA1c <7%)
* Microalbuminuria in the upper range of normal (> 150 <300 mg/24 h)

Exclusion Criteria:

* Pregnancy, lactation or women of childbearing age.
* Inability to stop treatment in place for a few days during the wash-out.
* Sitting diastolic blood pressure> 100 mmHg or systolic pressure> 170 at the end of the wash-out.
* History of hypertensive encephalopathy or cerebrovascular accident within 12 months prior.
* Secondary hypertension.
* Heart failure
* Acute myocardial infarction; angina pectoris
* Liver and kidney dysfunction
* Known hypersensitivity to ACE inhibitors
* All other physiological or pathological condition that the physician may affect the evaluation of the parameters under study or interfere with the proper conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Size of the reduction of urinary albumin in 24 hours to the various controls | After 12 weeks from the beginning

SECONDARY OUTCOMES:
1. Size of the reduction of mean 24-hour average daytime and nighttime average. 2. Size of the reduction of central blood pressure. 3. Magnitude of changes in plasma concentrations of angiotensin II, bradykinin and BNP after 24 weeks of treatment. | After 12 weeks from the beginning

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogari, MD, Study Director — University of Pavia
Locations (1):
- University of Pavia, Pavia, Italy